CLINICAL TRIAL: NCT03252691
Title: Study to Determine Incidence of Large Annular Defects And Measurement of Volume of Nucleus Removed in Primary Discectomy Patients
Brief Title: Incidence of Large Annular Defects in Primary Lumbar Discectomy Patients
Acronym: USLSI
Status: Withdrawn | Type: Observational
Why Stopped: Site closure and no patient enrolled
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: USCONTROL-USLSI-001
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Disc Herniation; Anular Tear of Lumbar Disc; Nucleus Pulp Hernia;Lumbosac
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lumbar discectomy study, collection and evaluation of incidence of large annular defects.

DETAILED DESCRIPTION:
This study is designed as a single-site prospective data collection. Measurements will be collected during 150 consecutive standard of care primary lumbar discectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18-75 years of age, and skeletally mature
2. Must have clinical and radiological evidence of primary lumbar disc herniation at one level of the lumbar spine between L3-S1.
3. Must be psychosocially, mentally and physically able to comply with protocol, post-operative management and follow-up care.
4. Subject must understand and sign the written Informed Consent.

Exclusion Criteria:

1. Prior surgery at the index lumbar vertebral level.
2. Subject requires spinal surgery other than a discectomy (with or without laminotomy) to treat leg/back pain
3. Morbid obesity (BMI ≥ 40 kg/m2)
4. Investigational drug or device use within 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty (150) subjects will participate in the study. Participants will be between 18 and 75 years of age. All subjects will have been diagnosed with primary lumbar disc herniation requiring surgical discectomy as per the opinion of the treating surgeon. All subjects who meet the inclusion criteria, do not meet any of the exclusion criteria, and who elect to participate and sign the informed consent will be included in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Incidence of large defects noted on primary lumbar discectomy procedure. | Intra-operatively
  Annular defect size will be measured intra-operatively.

SECONDARY OUTCOMES:
Quantify the amount of nuclear disc material removed during primary lumbar discectomy procedure. | Intra-operatively
  Amount of nucleus removed will be measured intra-operatively.
Verify access to annular defect with approved manual surgical instruments. | Intra-operatively
  Access to the annular defect will be evaluated intra-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Davis, MD, Principal Investigator — Laser Spine Institute
Locations (1):
- Laser Spine Institute, Tampa, Florida, United States